CLINICAL TRIAL: NCT02428556
Title: FDA "Breakthrough Drugs": A Randomized Trial Testing the Effect of Alternative Language on Public Perceptions
Brief Title: FDA "Breakthrough Drugs": A Trial Testing the Effect of Alternative Language on Public Perceptions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: STUDY00028203
Record Dates: First submitted 2015-02-09; First posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Prescription Drugs
Keywords: Decision making

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Facts only (Active Comparator): Scenario describes study results without "breakthrough" language, "promising" language, no cautions about conditional approval
  Interventions: Other: Facts only
- promising language (Active Comparator): study description describes drug as "promising"; no warning about conditional approval
  Interventions: Other: promising language
- breakthrough with "may" warning (Active Comparator): study describes drug as "breakthrough"; warning that continued approval may be contingent on subsequent verification of clinical benefit in confirmatory trials
  Interventions: Other: breakthrough with "may" warning
- breakthrough with "is" warning (Active Comparator): study describes drug as "breakthrough"; warning that continued approval may be contingent on subsequent verification of clinical benefit in confirmatory trials
  Interventions: Other: breakthrough with "is" warning
- breakthrough only (Experimental): Scenario describes study results with "breakthrough" language, no cautions about conditional approval
  Interventions: Other: breakthrough only

INTERVENTIONS:
Other: Facts only — Communicate basic information about breakthrough drugs provided in FDA press release without using Breakthrough label
  Arms: Facts only
Other: promising language — Communicate basic information about breakthrough drugs provided in FDA press release, using language commonly used by FDA in describing breakthrough drugs ("promising drug")
  Arms: promising language
Other: breakthrough only — Communicate basic information about breakthrough drugs provided in FDA press release using Breakthrough label (similar to information found in FDA press releases)
  Arms: breakthrough only
Other: breakthrough with "may" warning — Adding a tentative disclaimer (similar to that found on the FDA labels of some breakthrough designation drugs): "Continued approval for this indication may be contingent upon verification and description of clinical trial benefit in confirmatory trials"
  Arms: breakthrough with "may" warning
Other: breakthrough with "is" warning — Adding a more definitive disclaimer to minimize inaccurate inference from Breakthrough terminology: "Continued approval for this indication is contingent upon verification and description of clinical trial benefit in confirmatory trials."
  Arms: breakthrough with "is" warning

SUMMARY:
OBJECTIVE: To learn how people understand language used by the FDA to describe certain newly approved medications called "breakthrough" drugs.

BACKGROUND: FDA allows drugs to be designated as breakthrough if there is preliminary evidence that it may offer a substantial improvement over available therapies. But consumers (and prescribers) may mistake the word - which in this context means very preliminary promise and lots of uncertainty - to mean the drug is proven to be much more effective or much safer than existing drugs.

METHODS: Internet survey (with colleagues from Carnegie Mellon University) using Amazon Mechanical Turk - a web tool that recruits people willing to do surveys (https://www.mturk.com/mturk/welcome). Participants will be asked to read a short scenario about a new drug (facts are based on a real drug but the investigators use a fictional name) and answer questions about how well they think the drug works, how safe it is, etc. People will be randomized to one of 5 versions of the scenario differing in how explicitly they explain what "breakthrough" means. The information in the scenario is drawn from FDA's own press release about the drug.

DETAILED DESCRIPTION:
An online sample of 600 American participants was recruited from Amazon's Mechanical Turk. Respondents were randomly assigned to 5 conditions in which they read an excerpt from a news article describing a newly FDA-approved fictionalized breakthrough therapy, Zykanta, for treating metastatic lung cancer. Information on this fictionalized drug was drawn from a real-life breakthrough designated drug so as to be able to provide as accurate an example as possible with respect to inherent uncertainty in risk and benefit. Each condition communicated information about Zykanta with a greater or lesser degree of transparency regarding the contingent nature of a breakthrough approved drug. All conditions contained the same factual information about the risks and benefits of the drug. In the first condition - a Purely Factual condition - participants read a clear and concise technical definition of breakthrough therapy designation about a drug that was approved 4 months ahead of schedule, without seeing the term 'breakthrough' attached to the drug. This condition provides the basic risk-benefit information made available by the FDA without loaded terminology. In the second condition, the factual information was enhanced by describing the drug as "Promising" - the language the FDA uses in press releases about breakthrough drugs. This condition provides a more tempered label for this designation, but a label nonetheless. In the third condition, the factual information was enhanced by describing the drug as "Breakthrough." In the fourth condition, factual information about the drug was enhanced by describing the drug as "Breakthrough", but additionally contained a Tentative Disclaimer about the possible uncertainty surrounding the drug. This condition reflects the information found in the small print of the labeling of some breakthrough drugs. In the fifth condition, the factual drug information was enhanced by describing the drug as "Breakthrough", but contained a more Definitive Disclaimer about the uncertainty surrounding the drug and its need for further testing.

Measures To determine whether the term 'breakthrough' resulted in mistaken inference about its safety and effectiveness, all participants were asked to make a choice between a 'breakthrough drug' or a drug that met the definition of breakthrough without the explicit use of the word "breakthrough" in the description ("If you had a potentially deadly medical condition and could choose between 2 drugs recently approved by FDA, which would you choose? (1) 'Axabex, a "breakthrough" drug newly approved by the FDA' or (2) 'Hypapax, a drug that has shown some early promise in drug trials but which has not been shown to improve survival or disease-related symptoms'). All participants were asked whether they had heard the term "breakthrough drug" prior to being asked the question. All participants also provided a written definition of a breakthrough drug.

After reading the news excerpt on the fictional breakthrough drug in each of the 5 conditions, participants were surveyed on the safety and efficacy of the drug described in the news excerpt ("How safe is Zykanta compared to other drugs approved to treat metastatic lung cancer?", "How risky is Zykanta compared to other drugs approved to treat metastatic lung cancer?", "Has Zykanta been proven to save the lives of patients with metastatic lung cancer," "How effective do you think Zykanta is at treating metastatic lung cancer?" "If a patient with metastatic lung cancer started to take Zykanta, what do you think would happen to their tumor over the next 6 months?" and "How effective is Zykanta compared to other drugs approved to treat metastatic lung cancer?") and the strength of the scientific evidence that the drug helps metastatic lung cancer ("How strong is the scientific evidence that Zykanta helps patients with metastatic lung cancer?" and "If you were deciding to take Zykanta, would you feel confident making that decision given your current knowledge of the drug?"). We also asked about the likelihood of a symptom that was explicitly stated as a common symptom in the drug description ("If a patient with metastatic lung cancer started to take Zykanta, how likely is it that they would experience abdominal pain within 6 months?") and about their own anticipated behavior with respect to the drug ("If you were diagnosed with metastatic lung cancer, would you want to take Zykanta?" and "If a close friend or family member was diagnosed with metastatic lung cancer, would you want them to take Zykanta?"). Each response was measured on a 4 or 5-point Likert scale.

ELIGIBILITY:
Inclusion Criteria:

english speaking adult

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
effectiveness of zykanta | within 1 day
  After reading description of a trial for a hypothetical drug, participants will be asked:
  How effective do you / think Zykanta is at treating metastatic lung / cancer? Response will be choice of one of the following Not at all effective Somewhat effective Very effective Completely effective

SECONDARY OUTCOMES:
effect on tumor | within 1 day
  If a patient with / metastatic lung cancer started to take Zykanta, what do you think / would happen to their tumor over the next 6 / months
  Choices:
  * Nothing
  * Shrink a little
  * Shrink a lot
  * Go away completely
strength of scientific evidence | within 1 day
  How strong is the scientific / evidence that Zykanta helps patients with metastatic lung / cancer?
  Choices
  * Extremely weak
  * Weak
  * Strong
  * Extremely strong
Interest in taking | within 1 day
  If a close friend or / family member was diagnosed with metastatic lung cancer, / would you want them to take / Zykanta?
  Choices
  * Definitely not
  * probably not
  * probably yes
  * definitely yes